CLINICAL TRIAL: NCT02805296
Title: Intensive Phototherapy, Double vs. Single, in Treatment of Neonatal Hyperbilirubinemia Using LED
Brief Title: High Intensity Phototherapy: Double vs. Single
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: N-20140010
Record Dates: First submitted 2016-06-06; First posted 2016-06-20 (Estimated); Last update posted 2016-06-20 (Estimated); Status verified 2016-06

CONDITIONS: Hyperbilirubinemia
MeSH Terms: conditions — Hyperbilirubinemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Double light (Active Comparator): High-intensity phototherapy with blue LED light from above combined with a fiber optic, blue LED blanket from below.
  Intervention: Light irradiance: 66 µW/cm2/nm + 39 µW/cm2/nm
  Interventions: Other: Light irradiance
- Single light (Active Comparator): High-intensity phototherapy with blue LED light from above. Intervention: Light irradiance: 66 µW/cm2/nm
  Interventions: Other: Light irradiance

INTERVENTIONS:
Other: Light irradiance — Comparison of double vs. single phototherapy

SUMMARY:
Intensive phototherapy in form of double light is used worldwide in the treatment of severe neonatal hyperbilirubinemia. It has been debated if there is an upper limit on the efficiency of phototherapy. This study investigates whether double phototherapy reduces total serum bilirubin faster than single light during intensive phototherapy, using light emitting diodes, and whether there is an upper limit for the efficacy of phototherapy.

DETAILED DESCRIPTION:
Hyperbilirubinemia occurs in 60 - 80 % of newborns during the first days of life, among others because of immaturity of the enzyme uridin-glukuronosyl-transferase (UGT1A1) in the liver. In seldom cases with very high total serum bilirubin concentration (TsB), bilirubin can cross the blood-brain barrier and the deposition of unconjugated bilirubin in the central nervous system may cause acute bilirubin encephalopathy (ABE). This can progress to chronic bilirubin encephalopathy (CBE), a devastating condition, which unfortunately still occurs, even in industrialised countries.

Hyperbilirubinemia gets severe for 2 - 6 % of infants born at term or late preterm, which means, they need treatment to prevent ABE and the treatment of choice is phototherapy due to its efficacy and safety. Hereby bilirubin in the skin and plasma is converted to photobilirubins; they are water-soluble and can be excreted through the liver without conjugation. They are presumably non-toxic. In most departments, single phototherapy is first choice. To avoid the above-mentioned damaging condition, it is very important to optimize phototherapy.

Former fluorescent tubes were used as light source, but now light emission diodes (LED) are used.

This study investigates whether double phototherapy reduces total serum bilirubin faster than single light during intensive phototherapy, using LED, and whether there is an upper limit for the efficacy of phototherapy.

It is a prospective, randomised controlled study. The infants will be randomized to either 1: Conventional phototherapy with blue LED light from above and a distance from light source to mattress of 30 cm, giving a light irradiance of 66 µW/cm2/nm or 2: Conventional phototherapy combined with a light blanket (Bilisoft) with a light irradiance by the skin of 39 µW/cm2/nm. TsB will be measured at start and after 12 - and 24 h of treatment. Based on the calculation of strength 72 infants will be needed in this study. As statistical methods t-tests will be used and multiple linear regression models will be used to adjust for confounding.

ELIGIBILITY:
Inclusion Criteria:

* Otherwise healthy newborn infants with hyperbilirubinemia without signs of hemolytic disease
* gestational age ≥33 weeks
* birth weight ≥1800 g
* The infants should be treatable in a cradle

Exclusion Criteria:

* Infants fulfilling the indications for exchange transfusion or double phototherapy due to a very high initial or rapidly increasing TsB will not be enrolled.

Ages: 1 Day to 14 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 83 (Actual)
Dates: Start 2014-06; Primary Completion 2015-01 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Decrease in total serum bilirubin after 12- and 24 hours of phototherapy, measured in percent. | 12 and 24 Hours og phototherapy
  Total serum bilirubin will be measured at start of phototherapy, after 12 - and after 24 hours of phototherapy for both Groups. Primary outcome measure is, whether double phototherapy decreases total serum bilirubin faster than single phototherapy after 12- and/or after 24 hours of phototherapy.

SECONDARY OUTCOMES:
Whether total serum bilirubin continues to decrease measured in percent after 24 hours of high-intensity phototherapy | 24 Hours of phototherapy
  To figure out, whether there is an upper limit for the efficacy of phototherapy, i.e. a plateau above which total serum bilirubin does not decrease any further.

CONTACTS AND LOCATIONS:
Overall Officials: Mette L Roed, MD, Principal Investigator — Aalborg University Hospital

IPD SHARING:
Plan to Share IPD: No